CLINICAL TRIAL: NCT01028664
Title: Detection of IOP Fluctuation With SENSIMED Triggerfish in Patients With Glaucoma or Ocular Hypertension Treated With Diamox
Brief Title: Use of an Ocular Telemetry Sensor in Diamox Treated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Collaborators: Clinique de Montchoisi, Lausanne, Switzerland (Unknown)
Responsible Party: Prof. André Mermoud, Clinique de Montchoisi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09/05
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma and ocular hypertension patients
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glaucoma or ocular hypertension patients (Experimental)
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — 2-hour continuous IOP monitoring

SUMMARY:
A soft contact lens integrating a Sensor is placed on subjects with high intraocular pressure (IOP) after administration of an IOP-lowering drug to investigate the device's capacity to detect the induced IOP reduction.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of glaucoma or ocular hypertension
* IOP of ≥ 15 mmHg.
* Patients of either gender.
* Older than 18 years.
* Patients who accept signing an informed consent approved by the Ethics Committee.

Exclusion Criteria:

* Patients not able to understand the nature of the research
* Patients under tutorship
* Corneal abnormalities in both eyes
* Subjects with contraindications for wearing contact lenses
* History of ocular surgery within the last 3 months
* Known hypersensitivity to Diamox® or to any of its excipients
* Pregnancy and lactation
* Simultaneous participation in other clinical research
* Patients with evidence of ocular infection or inflammation
* History of renal or hepatic impairment, hypokalemia and hyponatremia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Detection of IOP reduction 2 hours after Diamox administration | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de Montchoisi, Centre du Glaucome, Lausanne, Switzerland